CLINICAL TRIAL: NCT02516475
Title: Effects of Zinc Supplementation on Weight, Body Mass Index (BMI), Waist Circumference, Fat Mass and Lean Mass, Apelin and Inflammatory Markers in Obese Individuals
Brief Title: Effects of Zinc Supplementation on Anthropometric Factors, Apelin and Inflammatory Markers in Obese Individuals
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 055570
Record Dates: First submitted 2015-07-30; First posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Zinc Sulfate; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zinc sulfate (Active Comparator): 1 zinc sulfate capsule for 15 weeks
  Interventions: Dietary Supplement: zinc sulfate
- starch (Placebo Comparator): 1 corn starch capsule for 15 weeks
  Interventions: Other: corn starch

INTERVENTIONS:
Dietary Supplement: zinc sulfate — 1 zinc sulfate capsule for 15 weeks
  Arms: zinc sulfate
Other: corn starch — 1 corn starch capsule for 15 weeks
  Other Names: placebo
  Arms: starch

SUMMARY:
To study the effects of zinc supplement on anthropometric factors, Apelin and inflammatory markers in obese individuals, 50 obes person who referred to Diet and Nutrition clinic of Shahid Beheshti University of Medical Sciences will be randomly allocated to receive 50 mg zinc capsules or placebos for 15 weeks; both groups will be advised to adherence the investigators' diet . At the first and the end of the intervention,weight, body mass index (BMI), waist circumference, fat mass and lean body mass, concentration of zinc, albumin, hs-CRP, TNF-α and plasma apelin will be assessed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 45 years
* Non-smoking
* Body Mass Index (BMI) more than 30

Exclusion Criteria:

* Pregnancy, lactation or menopause in women
* History of liver disease, kidney, thyroid, diabetes and other metabolic diseases
* Use of drugs interfering with lipid profile, blood-thinning drugs, beta-blockers
* Patients with immune deficiency
* Use of zinc, calcium and iron supplement in the last 2 months
* Use of weight loss medication or special diet
* Following program to lose weight in recent 2 months
* Recent surgery

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
weight | 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Azita Hekmatdoost, MD,PHD, Principal Investigator — National Nutrition and Food Technology Research Institute

REFERENCES:
- [Derived] Khorsandi H, Nikpayam O, Yousefi R, Parandoosh M, Hosseinzadeh N, Saidpour A, Ghorbani A. Zinc supplementation improves body weight management, inflammatory biomarkers and insulin resistance in individuals with obesity: a randomized, placebo-controlled, double-blind trial. Diabetol Metab Syndr. 2019 Dec 2;11:101. doi: 10.1186/s13098-019-0497-8. eCollection 2019. PMID 31827626